CLINICAL TRIAL: NCT06412822
Title: Neutrophil Extracellular Traps (NET's) in Prevalent Kidney Stone, Cross-section, Non-drug Clinical Study-Analysis of Biological Fluids (Residual Human Body Material (RHBM)): STONET's Project
Brief Title: Neutrophil Extracellular Traps (NET's) in Prevalent Kidney Stone
Status: Recruiting | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Agnieszka Pozdzik, Nephrologist, Brugmann University Hospital
Other Study IDs: STONET's
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * plasma sample
  * serum sample
  * total blood EDTA for DNA
  * urine samples: 24h collections, fasting urine and 2nd morning urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STONE group: Adult subjects with kidney stones disease
  Interventions: Other: Blood sampling; Other: Urine sampling
- NON STONE group: Control group: patients with acute and/or chronic kidney disease (CKD) without stones
  Interventions: Other: Blood sampling; Other: Urine sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling
Other: Urine sampling — Urine sampling

SUMMARY:
Neutrophils are first responders to any kind of threat the body faces: infection, severe trauma, cancer, surgery... They produce the cytokines, induct oxidative stress and de-granulate toxic proteins to kill pathogens. However the new mechanism related to the neutrophil extracellular traps release has been recognized as a new way of cell necrosis and has been called a NETosis.

NETosis is a hugely important new mechanism of human immune responses also described in various forms of acute kidney injury (ischemic, toxic, autoimmune). In certain kidney diseases, neutrophils release NETs and induce cell necrosis. Whether neutrophils die along with NET release, and if they do die, remains under study and is most likely context dependent. Extracellular traps (ETs) can be released also by macrophages. The ETs formation as well as macrophages extracellular traps (MET's) especially in kidney disease are cytotoxic and elicit inflammation, contributing to necro-inflammation of the early-injury phase of acute tubular necrosis in anti-neutrophil cytoplasmic antibody-related renal vasculitis, anti-glomerular basement membrane disease, lupus nephritis. Finally, acute kidney injury-related releases of dying renal cells or ETs promote organ injuries - for example, acute respiratory distress syndrome. According to the recent review the term 'NET formation' has been proposed as a better term to use instead of 'NETosis'. The formation of neutrophil extracellular traps (NETs) has been recently recognized as a unique modality of pathogen fixation (sticky extracellular chromatin) and pathogen killing (cytotoxic histones and proteases) during host immune responses, as well as collateral tissue damage.

Histones are potent mediators of injury in various cells. Indeed, extracellular histone induce microvascular endothelial cells and renal epithelial cells death in vitro, forms the pores that disrupt cell integrity and induce the cytolysis by their capacity of binding with membrane phospholipids and activation of inflammasome in the kidney leading to auto-entrainment of inflammation.

The activation of inflammation has been demonstrated in the experimental model of crystalline nephropathy related to the uncontrolled oxalate urinary excretion. Inhibition of inflammasome activation has been related with the preservation of kidney function. In patients with kidney stone disease the presence of crystals in the urine has been demonstrated to induce tubular epithelial cells injury that can theoretically trigger the NET's or MET's release and tissue inflammation.

NETs are now increasingly described as new targets for therapies, however largely under-estimated.

The role of release of ETs from neutrophils and macrophages during the kidney stone disease has never been studied in urine but the neutrophil extracellular trap (NET) formation-NETosis - was found significantly increased in the papillae of patients with brushite stones compared with CaOx stones.

The key objectives of this study are:

1. to assess NET/MET's excretion in the urine as a non-invasive method of NET/MET'osis measurement in patients with kidney diseases as a new biomarker of early stage of cells damages reflecting kidney injury occurring in patients with uncontrolled stones and other renal diseases;
2. to compare the NET/MET's concentrations in the urine with those in plasma

ELIGIBILITY:
Inclusion Criteria:

- Patients with acute and/or chronic kidney disease, with stones or without stones, ambulatory or hospitalized in CHU Brugmann Brugmann.

Exclusion Criteria:

* Malignancy or treatment for malignancy within 12 months prior to Screening with the exception of localized basal cell or squamous cell skin cancer. Note: Subjects whose malignancy is in remission and who are on a stable dose of chronic suppressive or maintenance therapy are not excluded.
* Psychological illness or condition, interfering with the patient's compliance or ability to understand the requirements of the study.
* Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute and/or chronic kidney disease, with stones or without stones, ambulatory or hospitalized in CHU Brugmann Brugmann.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neutrophil extracellular traps (NETs) excretion in 24h urine collection | 24 hours
  Assessment of NET excretion in 24h urine collection
Neutrophil extracellular traps (NETs) excretion in fasting urine | 24 hours
  Assessment of NET excretion in fasting urine
Neutrophil extracellular traps (NETs) excretion in 2e morning urine | 24 hours
  Assessment of NET excretion in 2e morning urine
Macrophages extracellular traps (MET's) excretion in 24h urine collection | 24 hours
  Assessment of MET's in 24h urine collection
Macrophages extracellular traps (MET's) excretion in fasting urine | 24 hours
  Assessment of MET's in fasting urine
Macrophages extracellular traps (MET's) excretion in 2e morning urine | 24 hours
  Assessment of MET's in 2e morning urine

SECONDARY OUTCOMES:
Neutrophil extracellular traps (NETs) plasma levels | 24 hours
  Neutrophil extracellular traps (NETs) plasma levels
Macrophages extracellular traps (MET's) plasma levels | 24 hours
  Macrophages extracellular traps (MET's) plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka POZDZIK, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No